CLINICAL TRIAL: NCT04836312
Title: A Soft Commitment Device to Encourage Intermittent Fasting in Patients With the Metabolic Syndrome
Brief Title: Intermittent Fasting Adherence and Self Tracking
Acronym: iFAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 844153
Record Dates: First submitted 2021-03-22; First posted 2021-04-08 (Actual); Results first posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-02

CONDITIONS: Hypertension; Obesity
MeSH Terms: conditions — Hypertension; Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attention Control (No Intervention): Patients will be instructed via text message and email to fast at least 16 hours per day every day. For the next 18 weeks, they will receive a daily text message via the Way to Health platform asking if they fasted for at least 16 hours over the past 24 hours. If they fail to respond, reminder text messages will be sent. Once per week, they will receive a text message asking them to weigh themselves and check their blood pressure, and reply with the results via text message
- Soft Commitment Device (Experimental): Patients randomized to the commitment device arm will be asked to visit the Way to Health platform. There, they will identify a support person, a family or friend who they speak to frequently and who is invested in their health. They will then complete a series of questions intended to create implementation intentions. Specifically, they will pick a time for their fast to begin each 24-hour period and a time for their fast to end. They will also develop strategies to deal with hunger arising during a fast period. After this process, they will sign a contract pledging to adhere to the 16:8 time-restricted feeding dietary pattern, and acknowledging that their support person will receive a copy of the contract and weekly updates about their adherence to the regimen.
  Interventions: Behavioral: Soft Commitment Device

INTERVENTIONS:
Behavioral: Soft Commitment Device — Patients randomized to the commitment device arm will be asked to visit the Way to Health platform. There, they will identify a support person, a family or friend who they speak to frequently and who is invested in their health. They will then complete a series of questions intended to create implementation intentions. Specifically, they will pick a time for their fast to begin each 24-hour period and a time for their fast to end. They will also develop strategies to deal with hunger arising during a fast period. After this process, they will sign a contract pledging to adhere to the 16:8 time-restricted feeding dietary pattern, and acknowledging that their support person will receive a copy of the contract and weekly updates about their adherence to the regimen.
  Arms: Soft Commitment Device

SUMMARY:
This pilot study will randomize 34 patients with hypertension and obesity to either time-restricted feeding alone or a commitment device to encourage time-restricted feeding, including a commitment pledge, involvement of a supportive partner, setting of implementation intentions, and multiple daily reminder text messages. The intervention will last 12 weeks, followed by a 6-week follow-up period. The primary outcome is adherence to the IF regimen, captured via daily text message, over 18 weeks

DETAILED DESCRIPTION:
1.1. Non-Pharmacologic Interventions to Improve Blood Pressure Control: Despite the wide availability of multiple classes of antihypertensive agents, compelling data that blood pressure (BP) lowering reduces mortality and cardiovascular events, and decades of public health campaigns, half of American adults with hypertension do not achieve adequate BP control. Randomized controlled trials of interventions to improve BP control in patients with hypertension have largely focused on home blood pressure monitoring, nurse- or pharmacist-lead education and medication titration, and/or financial incentives. Though many of these interventions improve short-term blood pressure control, they are cost-additive to health systems, post-intervention data is mixed, and none have been widely implemented.

Though consensus guidelines recommend dietary changes to improve hypertension control, with a particular recommendation in favor of the DASH (Dietary Approaches to Stop Hypertension) diet, very few U.S. patients adhere to this complex dietary pattern. The DASH diet reduced systolic BP (SBP) by 11 mmHg in randomized controlled trials in which participants were provided with food, and 4 mmHg in a study testing a 6-month, 18-visit intensive lifestyle intervention intended to promote the DASH diet; however, BP control was not sustained 12 months after the end of the intensive intervention.

1.2. Effect of Intermittent Fasting on Metabolic Parameters: In contrast to the DASH diet, intermittent fasting (IF) is a dietary pattern that emphasizes temporal restriction of caloric intake rather than restricting the number of calories and/or changing the types of foods eaten. The simplest and most popular variation of IF involves restricting caloric intake to an 8-hour period each day, and consuming no calories for the other 16 hours (so-called 16:8 time-restricted feeding). In animal studies, IF has been shown to activate cellular pathways with potential disease-modifying benefits in a number of conditions. In small human studies, IF is associated with a reduction in SBP by 5-10 mmHg, LDL cholesterol by ~8 mg/dl, and weight by ~ 3 kg, though none of the studies of a time-restricted feeding regimen included concurrent controls. Some patients report that IF is easier to initiate and maintain than other dietary patterns, though this has not been tested empirically.

1.3. Commitment Devices to Promote Healthy Behaviors: Commitment devices are centered in theoretical research that posits a planner-doer framework, wherein an individual can be conceptualized as dual sub-selves: The planner, who cares about long-term well-being; and the doer, who cares only for the present and prioritizes immediate payoffs. Conflict between the motivations and priorities of the planner and the doer sub-selves results in failure to follow-through with a plan when the moment to act arrives. Commitment devices are mechanisms by which the planner sub-self constrains the actions of their future doer sub-self by making certain choices more costly. Hard commitments impose a financial penalty for failing to follow through on the commitment, and soft commitments impose a psychological penalty. Hard commitments have been shown to change health behaviors, as in a study where smokers forfeited money deposited in a savings account if they failed to quit smoking after 6 months. However, monetary losses may not be attractive to many people, and effective soft commitment devices may be more appealing.

Pre-clinical research suggests that both intra- and interpersonal commitments might be useful components of a soft commitment device. Intrapersonal commitments have also been framed as implementation intentions, or specific plans as to where, how, and/or when an action will be taken. In small experiments, smokers who set a quit date were more likely to quit, and college students who set a date and time to visit a vaccination clinic were more likely to receive their vaccination. Interpersonal commitments leverage social networks, so that the penalty involves letting down a support partner. Involvement of social networks has been used to increase physical activity and improve control of weight and blood glucose in patients with obesity and diabetes. Social networks have been used explicitly within the context of commitment devices to encourage deposits in a savings account in a study of Chilean micro-entrepreneurs who either attended or did not attend a weekly peer support group meeting. Weight loss studies encouraging participants to exercise and change their eating behavior have employed commitment devices, including some that leveraged the involvement of family members or friends of the participant, with mixed results.

1.4 Rationale for the IFAST Study: The IF dietary pattern, though not inspired by behavioral economic concepts, is structured to take advantage of them and thus may be particularly amenable to a robust commitment device intervention. Changing one's eating patterns to a complex new diet is a cognitively intense process that requires active consideration of complex information multiple times per day, leading to cognitive overload and impaired decision-making. By contrast, IF, especially time-restricted feeding, is cognitively very simple. This simplicity may help participants avoid cognitive overload, initiate the dietary pattern and adhere over the long term.

This study seeks to test how a robust soft commitment device, incorporating both intra- and interpersonal commitments, affects uptake and adherence to an intermittent fasting dietary pattern, as compared with control, in patients with obesity and hypertension

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Body mass index > 30 kg/m2
* Systolic blood pressure > 150 mmHg
* Owns a smartphone or tablet operating the iOS or Android operating system

Exclusion Criteria:

* Unable or unwilling to provide informed consent, including but not limited to cognitive or language barriers (reading or comprehension)
* Type 1 diabetes
* Use of insulin or insulin secretagogues (sulfonylureas, metaglinides)
* Use of medications that require food intake
* Ongoing use of pharmacologic therapy for weight loss
* Self-reported eating disorder
* Other medical condition that could be harmed by intermittent fasting as judged by study physician
* Anticipated life expectancy less than 6 months
* Any other reason why it is not feasible to complete the entire 6-month study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-08-28 (Actual); Study Completion 2022-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh Patel, MD, MBA, MS, Principal Investigator — University of Pennsylvania; Alexander Fanaroff, MD, MHS, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fanaroff AC, Coratti S, Halaby R, Sanghavi M, O'Quinn RP, Krishnan S, Glassberg H, Bajaj A, Adusumalli S, Chokshi N, Patel MS. Feasibility and outcomes from using a commitment device and text message reminders to increase adherence to time-restricted eating: A randomized trial. Am Heart J. 2023 Apr;258:85-95. doi: 10.1016/j.ahj.2022.12.010. Epub 2023 Jan 11. PMID 36640862

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Attention Control | Soft Commitment Device
Started | 20 | 17
Completed | 20 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Attention Control | Soft Commitment Device | Total
Number analyzed (Participants) | 20 | 17 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (11.8) | 60.1 (10.3) | 60 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 8 | 22
  Male | 6 | 9 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 17 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 2 | 12
  White | 9 | 15 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 17 | 37

OUTCOME MEASURES:

1. Primary Outcome: Adherence to the Intermittent Fasting Regimen, Captured Via Daily Text Message, Over 18 Weeks, Expressed in Days Per Week
Description: Adherence to the IF regimen, captured via daily text message, over 18 weeks, expressed in days per week. This will measure adherence to the IF regimen throughout the 12 week intervention period and the 6 week follow-up period.
Time Frame: Weeks 1-18
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Attention Control | Soft Commitment Device
Number analyzed (Participants) | 20 | 17
days per week | 4.7 (1.9) | 5.4 (1.7)

2. Secondary Outcome: Adherence to the IF Regimen, Captured Via Daily Text Message, Over 12 Weeks, Expressed in Days Per Week
Description: Adherence to the IF regimen, captured via daily text message, over 12 weeks, expressed in days per week. This will measure adherence to the IF regimen for the 12 week intervention period only.
Time Frame: Weeks 1-12
Measure: Mean (Standard Deviation); unit: days per week
Arm/Group | Attention Control | Soft Commitment Device
Number analyzed (Participants) | 20 | 17
days per week | 5.0 (1.8) | 5.7 (1.6)

ADVERSE EVENTS:
Time Frame: 18 weeks
Arm/Group | Attention Control | Soft Commitment Device
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/17
Other Adverse Events (participants affected / at risk) | 0/20 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/12/NCT04836312/Prot_SAP_000.pdf